CLINICAL TRIAL: NCT06150196
Title: Comparison of Mindfulness-Wellness Class Versus Brain Health Education in Veterans With mTBI
Brief Title: Brain Health & Wellness Classes for Veterans With Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Bay Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-22-1-0820
Record Dates: First submitted 2023-10-12; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Brain Injury Traumatic Mild; Post-traumatic Stress Disorder
Keywords: Mindfulness; Mindfulness-based Stress Reduction; TBI; Anxiety; PTSD; Veteran
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Stress Reduction class (Experimental): Mindfulness-based Stress Reduction (MBSR) is a 9-week class that meets 2.5 hours/week and involves training in mindfulness (being present in the moment), meditation, and yoga. The MBSR course is taught by a certified MBSR instructor.
  Interventions: Behavioral: Mindfulness-based Stress Reduction class
- Brain Health Education Class (Active Comparator): the Brain Health Education Class is a 9-week class that meets 2.5 hours/week and involves lectures/discussion about how the brain works, how the brain ages, neuroplasticity, and other topics on the brain.
  Interventions: Behavioral: Brain Health Education class

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction class — 9-week standard Mindfulness-based Stress Reduction class training on mindfulness techniques, medication, and yoga
  Arms: Mindfulness-based Stress Reduction class
Behavioral: Brain Health Education class — 9-week Brain Health education class that involves lectures/discussion about how the brain works and recovers after brain injury
  Arms: Brain Health Education Class

SUMMARY:
This study is testing the usefulness of two types of Brain Health & Wellness classes for Veterans with a history of concussion to improve mental health.

DETAILED DESCRIPTION:
This is a pragmatic, randomized controlled trial of Mindfulness-based Stress Reduction (MBSR) in 120 Veterans with comorbid PTSD and chronic mTBI. Half of the participants are randomly assigned to MBSR and the other half, to a Brain Health education class, which serves as an active control group. A battery of standardized psychological and cognitive measures are administered prior to and following the class interventions to assess change in response to the intervention, with an additional 6-month follow-up assessment to test for lasting changes. The primary outcome measures include the Mayo-Portland Adaptability Inventory IV (functional outcome), PTSD Checklist (psychological outcome), and cognitive control test (cognitive outcome).

ELIGIBILITY:
Inclusion criteria:

* 18-75 years old
* chronic history (>6 months) of one or more mTBIs
* current diagnosis of PTSD
* at least one self-reported cognitive symptom

Exclusion criteria:

* no history of other neurologic disease (e.g., tumor, stroke, dementia, Parkinson's)
* no history of major brain surgery
* no history of moderate or severe TBI
* no active alcohol or drug dependence or abuse within previous 30 days
* no history of severe psychotic disorder (e.g., schizophrenia)
* no current suicidal ideation/risk
* no clinically severe medical illness requiring treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Mayo-Portland Adaptability Inventory | Within 2 weeks post-intervention
  Measure of Instrumental Activities of Daily Living with overall score of 0-111, with higher scores indicate greater impairment

CONTACTS AND LOCATIONS:
Locations (1):
- VA Northern California Health Care System, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: Undecided